CLINICAL TRIAL: NCT04507763
Title: Clinical Outcomes of Early Versus Delayed Management of Iraqi Patients With Ankylosing Spondylitis (AS) With Etanercept
Brief Title: Study To Evaluate The Impact Of Early Initiation Of Biological Treatment With Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801415
Record Dates: First submitted 2020-07-27; First posted 2020-08-11 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-09

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with ankylosing spondylitis: Iraqi patients diagnosed with ankylosing spondylitis that received Etanercept as treatment for disease
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Patients with ankylosing spondylitis as provided in real world practice
  Other Names: Enbrel

SUMMARY:
This study is to evaluate available data in Iraqi patients with ankylosing spondylitis on Enbrel treatment with regards to the impact of early treatment using data from the Baghdad Teaching Hospital registry

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed AS patients.

  * 18 years old
* Did not receive previous biological treatment for any reason

Exclusion Criteria:

* Patients previously or currently treated with other biological therapies.
* Use of etanercept for less than 1 year duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients data from local registry at the Baghdad Teaching Hospital
Sampling Method: Non-Probability Sample
Enrollment: 763 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1801415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of Iraq's participants aged greater than or equal to (>=) 18 years, who received etanercept for at least 1 year anytime from August 2012 through March 2020 for treatment of ankylosing spondylitis (AS) and met American College of Rheumatology/ European League Against Rheumatism (EULAR) 2019 criteria for AS were included in the study. Data were collected from dermatology center of Baghdad teaching hospital. Available data were evaluated in 2 months of this retrospective, observational study.
Groups:
- Etanercept: Participants received etanercept to treat AS for at least 1 year (anytime from August 2012 to March 2020) under standard real world clinical practice (In Iraq, the recommended dose of etanercept [Enbrel] is 25 milligrams [mg] administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly).Data of these participants were studied for 2 months in this retrospective, observational study.
Period: Overall Study
Arm/Group | Etanercept
Started | 763
Completed | 562
Not Completed | 201
Not completed — Participants did not meet entrance criteria | 201

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants whose data were included in the study for retrospective observation.
Groups:
- Etanercept: Participants received etanercept to treat AS for at least 1 year (anytime from August 2012 to March 2020) under standard real world clinical practice (In Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly).Data of these participants were studied for 2 months in this retrospective, observational study.
Arm/Group | Etanercept
Number analyzed (Participants) | 763
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 627
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education Level [Count of Participants; unit: Participants] — In this baseline measure, number of participants were classified according to their education level.
  Participants
    Primary education | 319
    Secondary education | 231
    Higher education | 213
Smoking Status [Count of Participants; unit: Participants] — In this baseline measure, number of participants were classified according to their smoking status as "Yes" or "No".
  Participants
    Yes | 389
    No | 374
Disease Duration [Mean (Standard Deviation); unit: Years] | 5.9 (6.1)
Current Steroid Therapy [Count of Participants; unit: Participants] — Population: In this baseline measure, number of participants who were on steroid therapy were reported.
  Participants | 614
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) [Mean (Standard Deviation); unit: Units on a scale] — BASDAI is a set of 6 questions to determine disease activity in participant with AS. Participants answered each 6 questions on a scale of 0 (no problem) to 10 (the worst problem). The BASDAI score is calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions (Q) 1-4. This score is then divided by 5. BASDAI score = (Q1 + Q2 + Q3+ Q4+ [Q5 + Q6/2])/5. BASDAI score ranges from 0 (best) to 10 (worst), where higher scores meant worse condition.
  Units on a scale | 8.1 (0.8)
Bath Ankylosing Spondylitis Functional Index (BASFI) [Mean (Standard Deviation); unit: Units on a scale] — BASFI is a set of 10 questions to determine degree of functional limitation in participants with AS. Participants answered each 10 questions on a scale of 0 (no functional impairment) to 10 (maximal impairment). BASFI total score was calculated as mean of scores from 10 questions. BASFI total score ranged from 0 (no functional impairment) to 10 (maximal impairment), where higher scores meant worse condition.
  Units on a scale | 7.7 (1.1)
Human Leukocyte Antigen B27 (HLA-B27) [Count of Participants; unit: Participants] — In this baseline measure, number of participants were classified according to presence of human leukocyte antigen B27 (HLA-B27) type as positive, negative and not done (if test not performed).
  Participants
    Positive | 242
    Negative | 167
    Not done | 354

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Total Score at Month 12
Description: BASFI is a set of 10 questions to determine degree of functional limitation in participants with AS. Participants answered each 10 questions on a scale of 0 (no functional impairment) to 10 (maximal impairment). BASFI total score was calculated as mean of scores from 10 questions. BASFI total score ranged from 0 (no functional impairment) to 10 (maximal impairment), where higher scores meant worse condition. In this outcome measure, participants were grouped on the basis of early and delayed referral to management of AS with etanercept treatment. Early referral was considered when participants were referred to management of AS in less than or equal to (<=) 1 year after diagnosis with AS. Participants with delayed referral to management of AS were divided into 3 groups: 1.1 to 5 years, 5.1 to 10 years and greater than (>) 10 years after diagnosis with AS.
Time Frame: Baseline, Month 12 [from the data retrieved and observed in 2 months of this study]
Population: Analysis population included all participants whose data were included in the study for retrospective observation. In this outcome measure, participants were grouped on the basis of early and delayed referral to management of AS with etanercept treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Etanercept: Participants With Early Referral (<=1 Year): Participants who were referred early (<=1 year after diagnosis with AS) for management of AS with etanercept treatment and received etanercept for at least 1 year (anytime from August 2012 to March 2020) under standard real world clinical practice (In Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly). Data of these participants were studied for 2 months in this retrospective, observational study.
- Etanercept: Participants With Delayed Referral (1.1 to 5 Years): Participants who were referred delayed (1.1 to 5 years after diagnosis with AS) for management of AS with etanercept treatment and received etanercept for at least 1 year (anytime from August 2012 to March 2020) under standard real world clinical practice (In Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly). Data of these participants were studied for 2 months in this retrospective, observational study.
- Etanercept: Participants With Delayed Referral (5.1 to 10 Years): Participants who were referred delayed (5.1 to 10 years after diagnosis with AS) for management of AS with etanercept treatment and received etanercept for at least 1 year (anytime from August 2012 to March 2020) under standard real world clinical practice (In Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly). Data of these participants were studied for 2 months in this retrospective, observational study.
- Etanercept: Participants With Delayed Referral (>10 Years): Participants who were referred delayed (>10 years after diagnosis with AS) for management of AS with etanercept treatment and received etanercept for at least 1 year (anytime from August 2012 to March 2020) under standard real world clinical practice (In Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly).. Data of these participants were studied for 2 months in this retrospective, observational study.
Arm/Group | Etanercept: Participants With Early Referral (<=1 Year) | Etanercept: Participants With Delayed Referral (1.1 to 5 Years) | Etanercept: Participants With Delayed Referral (5.1 to 10 Years) | Etanercept: Participants With Delayed Referral (>10 Years)
Number analyzed (Participants) | 239 | 209 | 138 | 177
Units on a scale
  Baseline | 7.75 (1.11) | 7.74 (1.11) | 7.72 (1.15) | 7.78 (1.13)
  Change from baseline at month 12 | -6.21 (1.557) | -5.44 (1.510) | -4.14 (1.697) | -4.04 (1.631)
Statistical Analysis 1: Comparison: Etanercept: Participants With Early Referral (<=1 Year); Change from Baseline at Month 12: For Early Referral; Test type: Other; p = 0.001, Regression, Logistic

2. Primary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score at Month 12
Description: BASDAI is a set of 6 questions to determine disease activity in participant with AS. Participants answered each 6 questions on a scale of 0 (no problem) to 10 (the worst problem). The BASDAI score is calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions (Q) 1-4. This score is then divided by 5. BASDAI score = (Q1 + Q2 + Q3+ Q4+ [Q5 + Q6/2])/5. BASDAI score ranges from 0 (best) to 10 (worst), where higher scores meant worse condition. In this outcome measure, participants were grouped on the basis of early and delayed referral to management of AS with etanercept treatment. Early referral was considered when participants were referred to management of AS in <= 1 year after diagnosis with AS. Participants with delayed referral to management of AS were divided into 3 groups: 1.1 to 5 years, 5.1 to 10 years and >10 years after diagnosis with AS.
Time Frame: Baseline, Month 12 [from the data retrieved and observed in 2 months of this study]
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept: Participants With Early Referral (<=1 Year) | Etanercept: Participants With Delayed Referral (1.1 to 5 Years) | Etanercept: Participants With Delayed Referral (5.1 to 10 Years) | Etanercept: Participants With Delayed Referral (>10 Years)
Number analyzed (Participants) | 239 | 209 | 138 | 177
Units on a scale
  Baseline | 8.32 (0.88) | 8.36 (0.47) | 8.46 (0.72) | 8.22 (0.86)
  Change from baseline at month 12 | -6.86 (1.550) | -6.05 (1.549) | -4.82 (1.782) | -4.4 (1.728)
Statistical Analysis 1: Comparison: Etanercept: Participants With Early Referral (<=1 Year); Change from Baseline at Month 12: For Early Referral; Test type: Other; p = 0.001, Regression, Logistic

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected for the study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not meet, hence adverse events were not collected and reported.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT04507763/Prot_SAP_000.pdf